CLINICAL TRIAL: NCT02438098
Title: Pharmacokinetics and Pharmacodynamics of Single Doses of Rivaroxaban in Obesity Patients Before and After Bariatric Surgery
Brief Title: Rivaroxaban in Bariatric Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 025/15
Record Dates: First submitted 2015-04-28; First posted 2015-05-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Prophylaxis of Venous Thromboembolism
Keywords: Rivaroxaban; Obesity; Bariatric surgery; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Obesity | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rivaroxaban arm (Other): Pharmacokinetics / Pharmacodynamics
  Interventions: Drug: Rivaroxaban 10 mg

INTERVENTIONS:
Drug: Rivaroxaban 10 mg — Patients receive the day before the surgical intervention the first dose of Rivaroxaban (10 mg) p.o. The second tablet Rivaroxaban is administered on the third postoperative day.

SUMMARY:
Until now there ist no systematic investigation of the pharmacokinetic parameters of Rivaroxaban in obese patient undergoing bariatric surgery. The aim of this study is to investigate the pharmacokinetic and pharmacodynamic parameters of rivaroxaban in obese patients before and after bariatric surgery.

Patients receive the day before the surgical intervention the first dose of Rivaroxaban (10mg). During the following 24 hours, 9 blood samples are taken.

The second tablet Rivaroxaban is administered on the third postoperative day, followed again by 9 blood samples during the next 24 hours.

All other blood samples are taken independent from this clinical trial as part of the standard medical treatment during the hospitalization. The hospital stay will not be extended by the study. The outpatient regular follow-up takes place one month after surgery and is combined with the last study visit.

DETAILED DESCRIPTION:
Background

The prevalence of obesity and morbid obesity is increasing worldwide and is becoming an increasing medical and socioeconomic burden. Bariatric surgery leads to the most sustained reduction of weight and associated co-morbidities. Obesity is a risk factor for the development of venous thromboembolism and the association between obesity and postoperative VTE is well established. The incidence of symptomatic DVT and PE ranges from 0%-5.4%, respectively 0%-6.4% and remains uncertain. Although the overall incidence seems to be low, VTE represents a significant cause of morbidity and mortality after surgery. Most postdischarge VTE events occur within the first 30 days after surgery and therefore extended chemoprophylaxis after hospital discharge is the standard of care and should be considered especially for patients classified to be at high risk for VTE.

Anticoagulants are recommended for the prevention of VTE, but there is no consensus regarding optimal method of prophylaxis. Routine perioperative use of drugs such as low-molecular weight heparins (LMWHs), intermittent pneumatic compression and early mobilization are currently the major accepted forms. However, there is currently no class I evidence to provide guidance regarding the type or dose of antithrombotic prophylaxis after bariatric surgery. For parenteral application there is for example limited evidence to guide dosing of thromboprophylaxis in morbid obesity and higher dosages are necessary, because impaired absorption after subcutaneous application.

The knowledge of the effect of extremely high body weight on pharmacokinetic and pharmacodynamics parameters after bariatric surgery especially for novel orally administered anticoagulants that target specific factors in the coagulation cascade is scarce. One promising therapeutic option is rivaroxaban (BAY 59-7939, Rivaroxaban), an orally administered direct factor Xa inhibitor that is approved for several indications in the field of prevention and treatment of thromboembolic disorders.

In several types of bariatric surgery procedures, such as sleeve gastrectomy, Roux-en-Y gastric bypass and biliopancreatic diversion different parts of gastrointestinal tract are bypassed or removed. This could affect the absorption of medications. Absorption of rivaroxaban is dependent on the site of drug release in the GI tract. In a study looking at administration of the crushed tablet via a tube, a 29% and 56% decrease in AUC and Cmax compared to an oral tablet was reported when rivaroxaban granulate is released in the proximal small intestine. The effect of altered anatomy due to RYGB on oral drug absorption and bioavailability is currently unknown. Previous studies focused on drugs like metformin, sertraline or tacrolimus, but they yielded conflicting results. In a case report by Mahlmann et al. the absorption of rivaroxaban was immediate and not significantly impaired by bariatric surgery of the upper GI tract. However, data from larger patient collectives are not available.

Rivaroxaban is already approved for VTE prophylaxis in orthopaedic patients. Up to now, there is no clinical data available regarding obese patients after bariatric surgery. To fill this gap, this phase 1 clinical trial was designed with a study design that allows for intra-patient comparison of the effect of the bariatric surgery regarding pharmacokinetic and pharmacodynamics analysis.

Rivaroxaban as an oral anticoagulant could be an attractive option for VTE prophylaxis compared to subcutaneous (LMWH) standard treatment after bariatric surgery. Especially high-risk patients (high BMI, a history of DVT, obesity hypoventilation syndrome, pulmonary hypertension, hormonal therapy, venous stasis disease, male gender, expected long operative time or open approach, where an extended duration of thromboprophylaxis after hospital discharge is recommended, an oral therapy would be attractive.

Until now there is no systematic investigation of pharmacokinetic parameters of rivaroxaban in obese patient undergoing bariatric surgery. This phase I clinical trial offers the unique opportunity to investigate PK/PD in morbidly obese patients pre and post bariatric surgery. The results of this trial will help to design larger trials in this particular patient population with the final goal of safe and efficient use of rivaroxaban in morbidly patients.

Objective

The aim of this study is to investigate the pharmacokinetic and pharmacodynamic parameters of rivaroxaban in obese patients before and after bariatric surgery.

Methods

Investigation of rivaroxaban AUC in bariatric.

ELIGIBILITY:
Inclusion Criteria:

* Patient with scheduled elective bariatric surgery : laparoscopic Roux-en-Y gastric bypass surgery or sleeve resection
* Patient aged 18 years and older
* BMI 35kg/m^2 and higher
* Women of child bearing age: willingness of using a double barrier contraception method during the study
* Informed Consent as documented by signature

Exclusion Criteria

* Intake of oral anticoagulants (phenprocoumon, acenocoumarol, dabigatran, etexilate, apixaban etc.) 4 weeks prior to inclusion in the study
* Application of parenteral anticoagulants (unfractionated heparin, low molecular weight heparins, heparin derivates (fondaparinux etc.) 4 weeks prior to inclusion in the study
* Pharmacologic platelet inhibition 4 weeks prior to inclusion in the study
* Known coagulation disorders (e.g. Willebrand's disease, haemophilia)
* Evidence for deep vein thrombosis or pulmonary embolism in the personal history or in the history of first degree relatives
* Medical condition that is associated with an increased risk for VTE, i.e. active cancer disease, lupus erythematodes chronic inflammatory bowel disease
* Active, clinically significant bleeding
* Congenital or acquired bleeding disorder
* Uncontrolled severe hypertension
* Active gastrointestinal disease that can potentially lead to bleeding disorder: oesophagitis, gastritis, gastroesophageal reflux disease, chronic inflammatory bowel disease
* Vascular retinopathy
* Bronchiectasis or history of pulmonary bleeding
* Prior stroke or TIA
* Hereditary galactose intolerance, Lapp lactase deficiency, glucose-lactose malabsorption
* Severe renal impairment with a creatinine clearance (GFR) of <30ml/min
* Positive pregnancy test, pregnancy or nursing women
* High risk of bleeding (e.g. active ulcerative gastrointestinal disease)
* Known intolerance of the study medication rivaroxaban
* Concomitant treatment with strong CYP3A4 inhibitors (e.g. ketoconazole, itraconazole, lopinavir, ritonavir, indinavir)
* Concomitant treatment with an P-glycoprotein inhibitor and weak or moderate CYP3A4 inhibitor (e.g. erythromycin, azithromycin, diltiazem, verapamil, quinidine, ranolazine, dronedarone, amiodarone, felodipine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Geometric mean ratio of rivaroxaban AUC (after surgery / before surgery) | 1 year

SECONDARY OUTCOMES:
AUC of rivaroxaban | 1 year
Cmax of rivaroxaban | 1 year
Tmax of rivaroxaban | 1 year
Prothrombin time (PT) | 1 year
Activated partial thromboplastin time (aPTT) | 1 year
Prothrombin fragment (F1+F2) | 1 year
Thrombin-antithrombin-complexes (TAT) | 1 year
D-Dimers | 1 year
Thrombin generation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dino Kroell, ME, Study Chair — University of Bern
Locations (1):
- Department of Visceral Surgery and Medicine, University Hospital Bern, Bern, Switzerland